CLINICAL TRIAL: NCT02101476
Title: A Randomized, Open Label,Prospective Study of the Analgesic Efficacy of Oral Xartemis Compared to Generic Oxycodone/APAP (Acetaminophen) in the Treatment of Moderate to Severe Post Operative Pain
Brief Title: An Open Label, Prospective Study of the Analgesic Efficacy of Oral Xartemis Compared to Generic Oxycodone/APAP( Acetaminophen) in the Treatment of Moderate to Severe Post Operative Pain.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lotus Clinical Research, LLC (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCR-MNK-01C
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Post Operative Pain
Keywords: Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percocet (Active Comparator): Oxycodone/APAP (acetaminophen)
  Interventions: Drug: Percocet
- Xartemis (Active Comparator)
  Interventions: Drug: Xartemis

INTERVENTIONS:
Drug: Percocet — 10mg/650mg
  Other Names: Oxycodone/APAP(acetaminophen)
  Arms: Percocet
Drug: Xartemis — 15mg/650mg
  Arms: Xartemis

SUMMARY:
The purpose of this study is to compare the analgesic efficacy of Xartemis 15mg/650mg by mouth every 12 hours for the management of acute moderate to severe post operative pain to generic Oxycodone/APAP(acetaminophen) (Percocet) 10mg/650mg by mouth every 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide written informed consent prior to enrollment
* Male or female and 18 years of age or older.
* Patients who are scheduled to undergo elective general surgery including, but not limited to the following surgical types:

  * Abdominal surgery
  * Orthopedic surgery
  * Spine surgery
  * Genitourinary surgery
* Patient classified as American Society of Anesthesiologists (ASA class I-III).
* Female subjects are eligible only if all of the following apply:

  * Not pregnant (subjects of child bearing potential must have a negative beta human chorionic gonadotropin (β-hCG) pregnancy test before surgery);
  * Not lactating;
  * Not planning to become pregnant within the duration of the study;
* Patients who are expected to have acute pain requiring oral opioid analgesics for at least 48 hours during the post operative period (either inpatient or outpatient).
* Patient must report a categorical pain rating of moderate to severe on a scale of none, mild, moderate, or severe prior to randomization.
* Patients who are willing and capable of understanding and cooperating with the requirements of the study.
* Patients able to understand and communicate in English.

Exclusion Criteria:

* Patients with a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation, safety, or conduct of the study such as but not limited to a history of severe renal or hepatic impairment, severe active hepatic disease, or any other clinically significant medical condition that may preclude safe study participation
* Patients who have a known severe allergy or hypersensitivity to opioid analgesics, anesthetics, APAP (acetaminophen.)
* Patients who have a history of intolerance to short term opioid use.
* Patients who have abused any prescription medication or alcohol within two years before the start of the study.
* Patients who require an additional scheduled surgical procedure within 48 hours of the surgery.
* Patients who have a history of seizures, or are currently taking anticonvulsants.
* Patients who have dysphagia and/or cannot swallow study medication whole.
* Patient who is unable to adequately communicate with study staff, properly give informed consent, or otherwise comply with study procedures.
* Patient who has participated in another clinical trial of an investigational drug or device within 30 days of screening visit or is schedule to receive an investigational product while participating in the study.

Post operative Exclusion Criteria at Randomization:

* Patients who are not awake, not breathing spontaneously, or have a respiratory insufficiency.
* Patients who are vomiting and not responsive to standard treatment
* Patients not able to answer questions and follow commands.
* Patients who have surgical complications that could compromise safety of the subject or confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Non Inferiority | 48 Hours
  To demonstrate the non inferiority of Xartemis 15mg/650mg by mouth every 12 hours for the management of acute post operative pain when compared to generic Oxycodone/APAP (acetaminophen) 10mg/650mg by mouth every 6 hours. The statistical comparison of interest will be the patient global assessment of analgesic effect administered at 48 hours after treatment initiation.

SECONDARY OUTCOMES:
Patient Global Assessment | 120 Hours
  To assess patient global assessments at 120 hours after treatment initiation for Xartemis 15mg/650mg by mouth every 12 hours compared to generic Oxycodone/APAP (acetaminophen) 10mg/650mg by mouth every 6 hours.

OTHER OUTCOMES:
Healthcare Professional Global Assessment | 48 Hours
  To assess healthcare professional global assessments at 48 hours and 120 hours after treatment initiation for Xartemis 15mg/650mg by mouth every 12 hours compared to generic Oxycodone/APAP (acetaminophen) 10mg/650mg by mouth every 6 hours.
Healthcare Professional Global Assessment | 120 Hours
  To assess healthcare professional global assessments at 48 hours and 120 hours after treatment initiation for Xartemis 15mg/650mg by mouth every 12 hours compared to generic Oxycodone/APAP (acetaminophen) 10mg/650mg by mouth every 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Singla, MD, Principal Investigator — Lotus Clinical Research, LLC
Locations (1):
- Lotus Clinical Resarch,LLC, Pasadena, California, United States